CLINICAL TRIAL: NCT00239928
Title: Long-Term Study For Pegaptanib Sodium In Patients With Subfoveal Choroidal Neovascularization Secondary To Age-Related Macular Degeneration (Extension Study From A5751010)
Brief Title: Clinical Study Of Pegaptanib Sodium (EYE001) For Wet-Type Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5751015
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Results first posted 2011-05-04 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2011-05

CONDITIONS: Macular Degeneration
Keywords: Long-Term Study For Pegaptanib Sodium In Patients With Subfoveal Choroidal Neovascularization Secondary To Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EYE001 (Experimental)
  Interventions: Drug: pegaptanib sodium

INTERVENTIONS:
Drug: pegaptanib sodium — 1 drop per dosed eye per protocol.

SUMMARY:
This study will examine the safety and efficacy of pegaptanib sodium in Japanese patients with wet-type age-related macular degeneration (AMD), who benefit further treatment and who want to continue the treatment after completion of the preceding study (A5751010).

ELIGIBILITY:
Inclusion Criteria:

* After completion of the preceding study (A5751010)

Exclusion Criteria:

* Serious heart, kidney and/or liver disease
* Diabetic retinopathy

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Japan (12):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Urayasu, Chiba
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Fukushima, Fukushima
  - Pfizer Investigational Site, Maebashi, Gunma
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Kyoto, Kyoto
  - Pfizer Investigational Site, Moriguchi, Osaka
  - Pfizer Investigational Site, Suita, Osaka
  - Pfizer Investigational Site, Ōtsu, Shiga
  - Pfizer Investigational Site, Chiyoda-ku, Tokyo
  - Pfizer Investigational Site, Shinjuku-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5751015&StudyName=Clinical%20Study%20Of%20EYE001%20For%20Wet-Type%20Age-Related%20Macular%20Degeneration

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects received a 0.3 mg or 1 mg/eye EYE001 (pegaptanib sodium) intravitreal injection every 6 weeks for 48 weeks in the preceding study A5751010 (NCT00150202)
Groups:
- EYE001: All subjects received a 0.3 mg/eye EYE001 intravitreal injection every 6 weeks from Week 54 up to Week 198.
Period: Overall Study
Arm/Group | EYE001
Started | 61
Completed | 51
Not Completed | 10
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 4
Not completed — Not need to continue study | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | EYE001
Number analyzed (Participants) | 61
Age, Customized [Number; unit: participants]
  < 18 years | 0
  18-64 years | 7
  >=65 years | 54
Age Continuous [Mean (Standard Deviation); unit: years] | 73.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 51
Region of Enrollment [Number; unit: participants]
  Japan | 61

OUTCOME MEASURES:

1. Secondary Outcome: Mean Change in Visual Acuity From Baseline of A5751010 (NCT00150202) to Each Observation Time Point
Description: Change: value at each observation time point minus value at baseline of A5751010 (NCT00150202).
  Visual acuity was measured as number of letters that the participants for this study could read in Early Treatment Diabetic Retinopathy Study (ETDRS) chart (eyesight-test chart).The best value in visual acuity using ETDRS chart is 85 and the worst value in visual acuity is 0.
Time Frame: Week 0 (baseline), every 18 weeks from Week 54 up to Week 198
Population: Among Intent-to-treat, 8 subjects who entered the current study 14 days or more after the completion of Study A5751010 were excluded from Intent-to-treat.
  Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | EYE001
Number analyzed (Participants) | 53
letters
  Week 54 | -3.2 (13.36)
  Week 72 | -3.3 (15.25)
  Week 90 | -4.7 (15.97)
  Week 108 | -8.6 (16.83)
  Week 126 | -8.6 (18.36)
  Week 144 | -10.1 (17.95)
  Week 162 | -10.4 (16.70)
  Week 180 | -10.4 (16.63)
  Week 198 | -10.3 (16.42)

2. Secondary Outcome: Mean Change in Visual Acuity From the Starting Point of Current Study to Each Observation Time Point
Description: Value at each observation time point minus value at Week 54 (initiation of current study).
  Visual acuity was measured as number of letters that the participants for this study could read in Early Treatment Diabetic Retinopathy Study (ETDRS) chart (eyesight-test chart).The best value in visual acuity using ETDRS chart is 85 and the worst value in visual acuity is 0.
Time Frame: Weeks 54, every 18 weeks from Week 54 up to Week 198
Population: Intent-to-treat, Among 61 subjects, for efficacy analyses, 1 subject had missing data at Week 72.
  Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | EYE001
Number analyzed (Participants) | 61
letters
  Week 72 | -0.1 (6.72)
  Week 90 | -1.4 (9.63)
  Week 108 | -4.8 (11.69)
  Week 126 | -4.5 (13.25)
  Week 144 | -6.1 (13.45)
  Week 162 | -6.3 (12.99)
  Week 180 | -6.3 (12.77)
  Week 198 | -6.2 (12.92)

3. Secondary Outcome: Number of Responders
Description: Responders defined as subjects having lost from baseline of A5751010 (NCT00150202) less than 15 letters of visual acuity; includes subjects with visual acuity gain.
Time Frame: Week 0 (baseline), every 18 weeks from Week 54 up to Week 198
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | EYE001
Number analyzed (Participants) | 53
participants
  Week 54 | 41
  Week 72 | 41
  Week 90 | 37
  Week 108 | 33
  Week 126 | 32
  Week 144 | 30
  Week 162 | 29
  Week 180 | 29
  Week 198 | 30

4. Secondary Outcome: Number of Subjects Gaining Vision From Baseline of A5751010 (NCT00150202)
Description: Subjects gaining vision: gain from baseline of more than 15 letters of visual acuity.
Time Frame: Week 0 (baseline), every 18 weeks from Week 54 up to Week 198
Population: Among Intent-to-treat, 8 subjects who entered the current study 14 days or more after the completion of Study A5751010 (NCT00150202) were excluded from Intent-to-treat.
  Last Observation Carried Forward
Measure: Number; unit: participants
Arm/Group | EYE001
Number analyzed (Participants) | 53
participants
  Week 54 | 4
  Week 72 | 7
  Week 90 | 7
  Week 108 | 6
  Week 126 | 6
  Week 144 | 5
  Week 162 | 6
  Week 180 | 5
  Week 198 | 5

5. Secondary Outcome: Number of Subjects Who Are Maintaining Vision From Baseline of A5751010 (NCT 00150202)
Description: Maintaining vision includes gaining 0 letter or more in visual acuity using Early Treatment Diabetic Retinopathy Study chart from baseline.
Time Frame: Week 0 (baseline), every 18 weeks from Week 54 up to Week 198
Population: Among Intent-to-treat, 8 subjects who entered the current study 14 days or more after the completion of Study A5751010 (NCT 00150202) were excluded from Intent-to-treat.
  Last Observation Carried Forward
Measure: Number; unit: participants
Arm/Group | EYE001
Number analyzed (Participants) | 53
participants
  Week 54 | 24
  Week 72 | 20
  Week 90 | 21
  Week 108 | 16
  Week 126 | 17
  Week 144 | 15
  Week 162 | 15
  Week 180 | 15
  Week 198 | 15

6. Secondary Outcome: Number of Subjects With Severe Vision Loss From Baseline of A5751010 (NCT 00150202)
Description: Subjects with severe vision loss: loss from baseline of >= 30 letters of visual acuity.
Time Frame: Week 0 (baseline), every 18 weeks from Week 54 up to Week 198
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | EYE001
Number analyzed (Participants) | 53
participants
  Week 54 | 0
  Week 72 | 1
  Week 90 | 4
  Week 108 | 7
  Week 126 | 6
  Week 144 | 7
  Week 162 | 6
  Week 180 | 7
  Week 198 | 7

7. Primary Outcome: Summary of Adverse Events
Description: Number of subjects with serious and non-serious adverse events: Subjects with ophthalmic adverse events: Subjects with severe adverse events that interferes significantly with subject's usual function: Subjects discontinued due to adverse events: Subjects with dose reduction or temporary discontinuation due to adverse events
Time Frame: Week 54 (initiation of A5751015 study) up to Week 198
Population: Intent-to-treat
Measure: Number; unit: participants
Arm/Group | EYE001
Number analyzed (Participants) | 61
participants
  Subjects with adverse events | 57
  Subjects with serious adverse events | 16
  Subjects with ophthalmic adverse event | 47
  Subjects with severe adverse events | 4
  Severe Myocardial Infarction | 1
  Severe Femur Fracture | 1
  Severe Gastric Cancer | 1
  Severe Pancreatic Carcinoma | 1
  Subjects discontinued due to adverse events | 4
  Subjects with dose reduction or temporary disconti | 4

ADVERSE EVENTS:
Arm/Group | EYE001
Serious Adverse Events (participants affected / at risk) | 16/61
Other Adverse Events (participants affected / at risk) | 43/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EYE001 (N=61)
Macular degeneration (Eye disorders) | 3 (3)
Angina pectoris (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Cataract traumatic (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Arteriosclerosis obliterans (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EYE001 (N=61)
Conjunctival hemorrhage (Eye disorders) | 14 (14)
Conjunctival hyperaemia (Eye disorders) | 10 (10)
Conjunctivitis (Eye disorders) | 8 (8)
Corneal erosion (Eye disorders) | 7 (7)
Eye pain (Eye disorders) | 9 (9)
Keratitis (Eye disorders) | 11 (11)
Visual acuity reduced (Eye disorders) | 7 (7)
Myodesopsia (Eye disorders) | 5 (5)
Punctate keratitis (Eye disorders) | 4 (4)
Retinal haemorrhage (Eye disorders) | 5 (5)
Nasopharyngitis (Infections and infestations) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days.Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites.Investigator may not disclose previously undisclosed confidential info other than study results.